CLINICAL TRIAL: NCT03192007
Title: Multi-Parametric MRI for Renal Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1610M96261
Record Dates: First submitted 2017-05-09; First posted 2017-06-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Renal Transplant Rejection
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Patients with Stable Renal Function: Patients will be given MRI
  Interventions: Device: Magnetic Resonance Imaging
- Patients with Worsening Renal Function due to complications: MRI
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Investigate anatomic and functional characteristics of transplant kidneys using MRI
  Other Names: MRI

SUMMARY:
The goals of this study are:

* To optimize and evaluate multiple kidney MRI methods; and
* To investigate the potential of MRI in the assessment of transplant kidney functions; To achieve these goals, we will perform pilot MRI studies with kidney transplant patients. We will study if MRI can reflect different levels of kidney function. The investigators will also evaluate if MRI can differentiate causes for declining kidney function. Finally, the investigators will explore how MRI measures changes before and after medical treatment for worsening kidney function.

You may be invited for MRI exams with different exam options. An MRI exam may use either of two types of MRI machines at the center for magnetic resonance research (CMRR): the 3 Tesla (3T) scanner and the 7 Tesla (7T) scanner. You may also be invited for a multi-session exam. A description of the MRI exam types with different exam options and the types of multi-session exams is provided later in this document.

DETAILED DESCRIPTION:
To achieve these goals, the investigators will perform pilot MRI studies with kidney transplant patients. The investigators will study if MRI can reflect different levels of kidney function. The investigators will also evaluate if MRI can differentiate causes for declining kidney function. Finally, the investigators will explore how MRI measures changes before and after medical treatment for worsening kidney function.

Subjects may be invited for MRI exams with different exam options. An MRI exam may use either of two types of MRI machines at the CMRR: the 3T scanner and the 7T scanner. Subjects may also be invited for a multi-session exam. A description of the MRI exam types with different exam options and the types of multi-session exams is provided later in this document.

ELIGIBILITY:
Inclusion Criteria:

* Renal Transplant Recipients
* Capable to consent
* English speaking
* For studies with patients with fast worsening renal function: An abrupt (within 48 h) reduction in kidney function currently defined as a percentage increase in serum creatinine of ≥50% (1.5-fold from baseline), or a reduction in urine output (documented oliguria of less than 0.5 mL/kg/h for more than 6 h).
* For patients with recovered renal allograft function after therapy: renal allograft function as measured by glomerular filtration rate (eGRF) has been recovered and stabilized above a clinical acceptable level, such as 15 ml/min/1.73 mm2.

Exclusion Criteria:

* On dialysis due to renal allograft failure
* Acute and chronic pulmonary disease
* Pregnancy as reported in CMRR Safety Screen
* Ferromagnetic implants
* Any foreign metal objects in the body
* History of shrapnel or shot gun injury
* Cardiac pacemakers
* Defibrillator
* Neuronal stimulator
* Magnetic aneurysm clip
* Large tattoos on the abdomen or the brain and neck, as determined by CMRR Safety Officer
* Hip replacement
* Too large to fit in the magnet (BMI >= 40, approx.)
* Severe claustrophobia

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The proposed studies are pilot studies to obtain preliminary data for the development of hypotheses and estimate the power for future large-scale studies. To accomplish the objectives of the proposed pilot studies, we will enroll a total of 140 renal transplant patients. Based on our previous experience, there will be about 20% patients who may withdraw after informed consent. Equal number of male and female subjects will be recruited for each patient group. In addition, the age of patients will be matched or ensured insignificant across the groups of the study objectives.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2027-07-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Anatomic and functional MRI characteristics in transplant kidneys with stable renal function | Baseline
  Investigate the correlations between anatomic and functional characteristics by MRI and the level of transplant renal function

SECONDARY OUTCOMES:
Anatomic and functional MRI characteristics of transplant kidneys with transplant complications | Baseline
  Investigate the anatomic and functional MRI characteristics of transplant kidneys with transplant complications with comparisons with those from transplant kidneys having stable renal function

CONTACTS AND LOCATIONS:
Locations (1):
- CMMR, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No